CLINICAL TRIAL: NCT01629264
Title: Influence of Pregnancy-related Hormonal Fluctuations on Corneal Biomechanics in Humans
Brief Title: The Influence of Hormonal Changes During Pregnancy on Corneal Biomechanics in Humans
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Farhad Hafezi, Professor and Chairman of Ophthalmology, University Hospital, Geneva
Other Study IDs: CER-11-180; GE-OPHT-2012-1 (Other: University of Geneva, Switzerland)
Record Dates: First submitted 2012-06-24; First posted 2012-06-27 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Pregnancy
Keywords: Cornea; biomechanics; pregnancy; keratoconus; refractive surgery
MeSH Terms: conditions — Corneal Diseases; Keratoconus | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Ocular Response Analyzer — To measure corneal biomechanics, specifically corneal hysteresis (CH) and the Corneal Resistance Factor (CRF). The devise measures in a non-contact manner, by analyzing the deformation of the cornea upon a defined pulse of air.
  Other Names: ORA
Device: Scheimpflug measurement — A Scheimpflug camera will be used in a non-contact manner to assess topographical data from the anterior and posterior corneal surface as well as detailed data on corneal thickness.
  Other Names: Pentacam
Other: Blood sample — A blood sample will be taken at 6 months after surgery to determine the levels of several hormones. The blood needed to détermine hormone levels during pregnancy will be acquired during the routine examinations that are performed during pregnancy. Here, blood is taken routinely and an additional volume is taken for the purpose of this study.

SUMMARY:
The intraocular pressure in the human bulbus requires that the "wall" of the eye shows a certain (bio)mechanical strength. The human cornea represents the anterior portion of this wall. Since several years, there is a growing interest in the ophthalmological community for identifying factors modulating the biomechanical stability of the human cornea. Reasons are twofold: advances in keratoconus research and the increasing numbers of refractive laser surgery procedures with (correspondingly) increasing numbers of complications due to non-respecting the limits of corneal biomechanics.

There is evidence that oestrogen, but also thyroïd hormone changes have a major impact on corneal biomechanics. A number of recent observational studies have reported on keratoconus and refractive laser surgery patients with decompensating biomechanics during pregnancy.

Both hormones also show physiological changes during pregnancy and little is known about the impact of these physiological changes on the human cornea.

The aim of this study is to establish baseline values for physiological changes in the human cornea during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Pregnancy confirmed by echography
* Before gestation week 14

Exclusion Criteria:

* Pre-existing corneal disease
* Previous eye surgery
* Inability to understand the nature of the study
* Patient with legal guardian

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women at the Dept. of Gynecology and Obstetrics of the University Hospital of Geneva
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Correlate oestradiol and TSH plasma changes with changes in corneal CRF and CH and topographical changes | 15 months
  3 examinations during pregnancy (gestation week 10-14, 20-26, and 36-40) and one visit at 6 months after pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Hafezi, MDPhD, Principal Investigator — University Hospital, Geneva
Locations (1):
- University Hospital Geneva, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gatzioufas Z, Thanos S. Acute keratoconus induced by hypothyroxinemia during pregnancy. J Endocrinol Invest. 2008 Mar;31(3):262-6. doi: 10.1007/BF03345600. PMID 18401210
- [Background] Giuffre G, Di Rosa L, Fiorino F, Bubella DM, Lodato G. Variations in central corneal thickness during the menstrual cycle in women. Cornea. 2007 Feb;26(2):144-6. doi: 10.1097/01.ico.0000244873.08127.3c. PMID 17251801
- [Background] Hafezi F, Iseli HP. Pregnancy-related exacerbation of iatrogenic keratectasia despite corneal collagen crosslinking. J Cataract Refract Surg. 2008 Jul;34(7):1219-21. doi: 10.1016/j.jcrs.2008.02.036. PMID 18571094
- [Background] Padmanabhan P, Radhakrishnan A, Natarajan R. Pregnancy-triggered iatrogenic (post-laser in situ keratomileusis) corneal ectasia--a case report. Cornea. 2010 May;29(5):569-72. doi: 10.1097/ICO.0b013e3181bd9f2d. PMID 20335804
- [Background] Spoerl E, Zubaty V, Raiskup-Wolf F, Pillunat LE. Oestrogen-induced changes in biomechanics in the cornea as a possible reason for keratectasia. Br J Ophthalmol. 2007 Nov;91(11):1547-50. doi: 10.1136/bjo.2007.124388. Epub 2007 Jun 25. PMID 17591666
- [Background] Suzuki T, Kinoshita Y, Tachibana M, Matsushima Y, Kobayashi Y, Adachi W, Sotozono C, Kinoshita S. Expression of sex steroid hormone receptors in human cornea. Curr Eye Res. 2001 Jan;22(1):28-33. doi: 10.1076/ceyr.22.1.28.6980. PMID 11402376
- [Background] Spoerl E, Zubaty V, Terai N, Pillunat LE, Raiskup F. Influence of high-dose cortisol on the biomechanics of incubated porcine corneal strips. J Refract Surg. 2009 Sep;25(9):S794-8. doi: 10.3928/1081597X-20090813-06. PMID 19772253